CLINICAL TRIAL: NCT03983902
Title: The Effect of Placental Transfusion Methods on the Potentially Transfusion Levels of Endothelial Progenitor Cell and CD34+ Hematopoietic Stem Cell
Brief Title: Placental Transfusion Methods and Stem Cells
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Emel Okulu,MD, Principal Investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ankara University-03
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Placental Transfusion; Stem Cells
Keywords: stem cell; newborn; endothelial progenitor cell; CD34+ hematopoietic stem cell; delayed cord clamping; umbilical cord milking; immediate cord clamping
MeSH Terms: conditions — Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delayed cord clamping (Active Comparator): Delayed cord clamping
  Interventions: Procedure: Delayed cord clamping
- Umbilical cord milking (Active Comparator): Umbilical cord clamping
  Interventions: Procedure: Umbilical cord milking
- Immediate cord clamping (Active Comparator): Immediate cord clamping
  Interventions: Procedure: Immediate cord clamping

INTERVENTIONS:
Procedure: Delayed cord clamping — Delayed cord clamping will occur for up to 2 minutes.
  Arms: Delayed cord clamping
Procedure: Umbilical cord milking — Umbilical cord milking will occur milking of the 30 cm of the cord from placental site to baby, at a speed of 5 cm/second, 3 times in preterm newborns, 4 times in term newborns.
  Arms: Umbilical cord milking
Procedure: Immediate cord clamping — Immediate cord clamping will occur in 20 seconds after birth.
  Arms: Immediate cord clamping

SUMMARY:
To measure the levels of endothelial progenitor cells and CD34+ hematopoietic stem cells levels, and placental residual volume by delayed cord clamping, umbilical cord milking or immediate cord clamping in newborns at different gestational weeks.

DETAILED DESCRIPTION:
Umbilical cord blood is a rich source of stem cells. Placental transfusion is the transfer of the placental blood to the baby until the cord clamped during the birth. Placental transfusion can be accomplished by delayed cord clamping or umbilical cord milking.

One group will receive 2 minutes of delayed cord clamping, the second group will receive umbilical cord milking and the third group will receive immediate cord clamping. Following the cord clamping, the blood samples will be taken from the placental site of the umbilical cord to measure the stem cells from all subjects and placental residual volume will be measured.

Delivery room conditions, hospitalization (if needed), short-term outcome during hospitalization, prematurity related morbidities (if baby is preterm) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

Born at 24 weeks to 42 weeks infants

Exclusion Criteria:

Without parental consent, known congenital anomalies

Max Age: 3 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
The levels of stem cells | 18-months
  Measurement of the levels of endothelial progenitor cells and CD34+ hematopoietic stem cells

SECONDARY OUTCOMES:
Placental residual volume | 18-months
  The placental residual volume by delayed cord clamping, umbilical cord milking or immediate cord clamping

CONTACTS AND LOCATIONS:
Overall Officials: Emel Okulu, MD, Principal Investigator — Ankara University

IPD SHARING:
Plan to Share IPD: No